CLINICAL TRIAL: NCT07367074
Title: Effect of an Educational Intervention on Sexual Function and Therapeutic Adherence in Women With Breast Cancer
Brief Title: Effect of an Educational Intervention in Women With Breast Cancer (EDU-INT-BC)
Acronym: EDU-INT-BC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituts Supérieurs des Professions Infirmières et Techniques de Santé, Morocco (Other)
Responsible Party: Principal Investigator, LAAMARI Safa, Master's student in advanced practices in oncology and palliative care, Instituts Supérieurs des Professions Infirmières et Techniques de Santé, Morocco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ISPITS-PAOSP-EDU-INT-BC-2025
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female NOS
Keywords: Breast cancer; Educational intervention; Sexual function; Therapeutic adherence
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This is a single-group interventional study with a pre-post design, in which all participants receive the same educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention Arm (Experimental): Participants assigned to this arm will receive a structured educational intervention focusing on breast cancer, treatment-related side effects, sexual health, and therapeutic adherence. The intervention consists of two educational sessions of two hours each, followed by follow-up support via WhatsApp. Outcomes will be assessed before the intervention and two months after its implementation.
  Interventions: Behavioral: Therapeutic Education Program for Women With Breast Cancer

INTERVENTIONS:
Behavioral: Therapeutic Education Program for Women With Breast Cancer — This intervention will consist of a structured therapeutic education program designed for women with breast cancer. The program will focus on disease-related information, treatment modalities and their associated side effects, sexual function, and strategies to improve therapeutic adherence.
  The intervention will include two face-to-face educational sessions, each lasting two hours, delivered by a midwife enrolled in the final semester of a Master's program in advanced practices in oncology and Palliatives Cares, followed by supportive follow-up via WhatsApp to reinforce key messages and address participants' concerns.
  The educational content will be adapted to participants' needs and health literacy levels. Outcomes related to sexual function and treatment adherence will be assessed before the intervention and two months after its implementation.

SUMMARY:
This study aims to evaluate the effect of an educational intervention on sexual function and therapeutic adherence among women with breast cancer followed in the medical oncology department of Ibn Tofail Hospital, affiliated with Mohammed VI University Hospital Center in Marrakech.

Participants will receive a structured therapeutic education program focusing on breast cancer, available treatments and their potential side effects, as well as treatment adherence and its prognostic significance. Educational sessions will be complemented by patient follow-up to reinforce key messages and support adherence.

The study will assess changes in sexual function and therapeutic adherence before and after the educational intervention.

DETAILED DESCRIPTION:
This is an interventional study without a control group aiming to evaluate the effect of an educational intervention on sexual function and therapeutic adherence among women with breast cancer followed in the medical oncology department of Ibn Tofail Hospital, affiliated with the Mohammed VI University Hospital Center (CHU) in Marrakech.

Methodology: Participants will be recruited among women aged over 18 years, diagnosed with breast cancer, receiving oral anticancer treatment, and willing to participate in the study. Sociodemographic and clinical data will be collected through interviews with the participants and by reviewing their medical records.

Intervention: The therapeutic education program will consist of two sessions conducted by a midwife experienced in breast and cervical cancer screening, enrolled in the final semester of the Master's program in Advanced Practice in Oncology and Palliative Care at ISPITS Marrakech. The sessions will address topics such as breast cancer, available treatments and their role, treatment-related effects on sexual function, as well as the importance of therapeutic adherence and behavioral coping strategies.

Evaluations: Outcomes will be assessed using validated questionnaires to evaluate sexual function and therapeutic adherence. The questionnaires will be administered before the intervention and two months after the educational intervention in order to assess changes in sexual function and therapeutic adherence among participants.

Ethical Considerations: The study will comply with all ethical principles, including obtaining informed consent and ensuring the participants' right to withdraw from the study at any time. The intervention has already received approval from the ethics committee and will also be approved by a research professor and a permanent faculty member trained in therapeutic education at ISPITS, as well as by a medical oncology professor at Mohammed VI University Hospital Center in Marrakech, prior to its implementation.

Data Analysis: Data will be analyzed using SPSS software. For variables not following a normal distribution, non-parametric statistical tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older.
* Diagnosed with breast cancer.
* Receiving oral anticancer treatment.
* Willing to participate in the study.
* Able to attend the educational sessions.
* Having access to a mobile phone (smartphone).

Exclusion Criteria:

* Women with communication disorders.
* Women with severe psychiatric disorders that will interfere with participation in the educational intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will be restricted to women diagnosed with breast cancer.
Enrollment: 65 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Function Score (FSFI) | Baseline and 2 months after the intervention
  Sexual function will be assessed using the Female Sexual Function Index (FSFI), a validated questionnaire with a total score ranging from 2 to 36, where higher scores indicate better sexual function.
  The primary outcome will be the change in the total FSFI score between baseline and two months after the educational intervention.

SECONDARY OUTCOMES:
Change in Therapeutic Adherence Score (ARMS-12) | Baseline and 2 months after the intervention
  Therapeutic adherence will be assessed using the Adherence to Refills and Medications Scale (ARMS-12), a validated questionnaire with a total score ranging from 12 to 48, where lower scores indicate better medication adherence.
  The secondary outcome will be the change in the total ARMS-12 score between baseline and two months after the educational intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology Department, Ibn Tofail Hospital, Mohammed VI University Hospital Center, Marrakesh, Marrakech-Safi, Morocco

IPD SHARING:
Plan to Share IPD: No